CLINICAL TRIAL: NCT04898855
Title: Programa Online De Intervenção Cognitivo-Comportamental Para O Tratamento Da Insónia Em Sobreviventes Oncológicos
Brief Title: Internet-delivered Cognitive-Behavioral Intervention for Insomniac Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Portuguese Cancer League (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Maria Inês Clara, PhD candidate, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020.05728.BD
Record Dates: First submitted 2021-05-12; First posted 2021-05-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Insomnia; Cancer; Cancer Survivors
Keywords: insomnia; cancer; CBTI; digital CBT-I; internet intervention; cancer survivors
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OncoSleep intervention (internet-delivered cognitive-behavioral treatment for insomnia) (Experimental): Participants assigned to the experimental group receive immediate access to the OncoSleep program, a web-based self-guided cognitive-behavioral intervention for insomnia consisting of 6 weekly sessions. A certified psychologist will monitor the participant's progress and provide feedback.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- waitlist control (No Intervention): Participants assigned to the waitlist control group receive access to the OncoSleep program after 8 weeks.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Treatment includes sleep hygiene, sleep restriction, stimulus control, and cognitive therapy.
  Other Names: OncoSleep
  Arms: OncoSleep intervention (internet-delivered cognitive-behavioral treatment for insomnia)

SUMMARY:
The main purpose of this study is to determine the treatment effects and acceptability of an internet-based cognitive-behavioral therapy intervention to improve the sleep of Portuguese cancer survivors with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Provided informed consent
* Ability to read and write in Portuguese
* Ability to use a computer and/or smartphone, and the internet
* History of cancer
* Having completed primary cancer treatment (survivors who are on hormone and/or other long-term maintenance therapy agencies are eligible to participate)
* Subclinical or significant symptoms of insomnia (ISI scores>=8)
* Ongoing sleep medication accepted if the dosage has been stable during the last 4 weeks

Exclusion Criteria:

* Age ≤ 18 years
* Another unstable condition (e.g., sleep, psychiatric or medical condition)
* Pregnancy or breastfeeding
* Concurrent CBT-I
* Habitual night shift, or rotating shift-workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-08-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | Changes from baseline to post-intervention (8 weeks after randomization)
  Insomnia Severity Index: validated questionnaire among cancer survivors; a 7-item scale with total scores between 0 and 28 where higher scores indicate greater severity

SECONDARY OUTCOMES:
Anxiety | Changes from baseline to post-intervention (8 weeks after randomization)
  Hospital Anxiety and Depression Scale (total subscale 0-21, higher scores denote highest anxiety level)
Depression | Changes from baseline to post-intervention (8 weeks after randomization)
  Hospital Anxiety and Depression Scale (total subscale 0-21, higher scores denote highest depression level)
Health-related quality of life | Changes from baseline to post-intervention (8 weeks after randomization)
  European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30; World Health Organization Quality of Life - Brief (overall scores 0-100, higher scores indicate higher quality of life)
Cancer-related fatigue | Changes from baseline to post-intervention (8 weeks after randomization)
  Multidimensional Fatigue Symptom Inventory-Short Form (overall score -24-96, higher scores denote higher levels of cancer-related fatigue)
Sleep efficiency | Changes from baseline to post-intervention (8 weeks after randomization)
  Sleep Diary
Total sleep time | Changes from baseline to post-intervention (8 weeks after randomization)
  Sleep Diary
Sleep onset latency | Changes from baseline to post-intervention (8 weeks after randomization)
  Sleep Diary
Number of nocturnal awakenings | Changes from baseline to post-intervention (8 weeks after randomization)
  Sleep Diary
Wake after sleep onset | Changes from baseline to post-intervention (8 weeks after randomization)
  Sleep Diary

OTHER OUTCOMES:
Insomnia Disorder remission (score&lt;8) and response (change ≥8) on the ISI | Post-intervention (8 weeks after randomization)
  Overall score 0-28 interpreted as follows: 0-7 absence of insomnia; 8-14 sub-threshold insomnia; 15-21 moderate insomnia; 22-28 severe insomnia
Acceptability | Post-intervention (8 weeks after randomization)
  Self-report scales of satisfaction, adherence and perceived helpfulness rated on 4-point Likert scales adapted from Manber et al. (2011)
Adherence | Post-intervention (8 weeks after randomization)
  Computed as the number of modules completed
Usability | Post-intervention (8 weeks after randomization)
  User Experience Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Clara MI, van Straten A, Savard J, Canavarro MC, Allen Gomes A. Web-based cognitive-behavioral therapy for insomnia in cancer survivors: The OncoSleep randomized trial. Sleep Med. 2025 May;129:67-74. doi: 10.1016/j.sleep.2025.02.021. Epub 2025 Feb 18. PMID 39987779
- See also: OncoSleep website — https://oncosleep.com/